CLINICAL TRIAL: NCT00171171
Title: A Study of Efficacy and Safety of Long-term Treatment With Deferasirox in Patients With Beta-thalassemia and Transfusional Hemosiderosis
Brief Title: A Study of Long-term Treatment With Deferasirox in Patients With Beta-thalassemia and Transfusional Hemosiderosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2402
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-11

CONDITIONS: Beta-Thalassemia; Hemosiderosis
Keywords: Thalassemia (beta-thal. major); Transfusional hemosiderosis; Deferasirox; Beta-thalassemia major patients; Unable to be chelated with deferoxamine or deferiprone
MeSH Terms: conditions — beta-Thalassemia; Hemosiderosis; Thalassemia | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox

SUMMARY:
Because patients with beta-thalassemia are unable to actively eliminate iron from the body, toxic and eventually lethal levels of iron can accumulate as a result of repeated blood transfusions. This study will evaluate the efficacy, safety and tolerability of deferasirox.

ELIGIBILITY:
Inclusion Criteria:

* Beta-thalassemia outpatients with transfusional hemosiderosis and unable to be chelated with deferoxamine (DFO) due to DFO being contra-indicated and/or due to documented unacceptable toxicity of DFO or documented poor response to DFO despite proper compliance, or documented non-compliance to DFO, with serum ferritin ≥ 500 ng/ml and LIC ≥ 2 mg/Fe/g dw liver
* Beta-thalassemia outpatients with transfusional hemosiderosis treated with deferiprone

Exclusion Criteria:

* Means levels of ALT > 300 U/L
* Serum creatinine above upper limit of normal
* Active hepatitis C or chronic hepatitis B receiving specific treatment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-05; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Liver Iron Concentration (as measured by biopsy) | at baseline and after 1 yeor of ICL670 treatment

SECONDARY OUTCOMES:
Iron balance, i.e. Total Body Iron Excretion (based on the iron influx as determined by the amount of red cells transfused and the change in total body iron (TBI) stores) | after 1 year of ICL670 treatment
Putative surrogate markers such as serum ferritin serum iron, serum transferrin and transferrin saturation | monthly assessments for 1 year
Adverse events | during 1 year ICL670 treatment
hematology and biochemistry, urinalysis | monthly assessments for 1 year ICL670 treatment
ECG and Echocardiography | 6-monthly for 1 year ICL670 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ali Taher, Ass.Prof., Principal Investigator — American University of Beirut Medical Center
Locations (5):
- Novartis Investigative Site, Cairo, Egypt
- Ali Taher, Beirut, Lebanon
- Novartis Investigative Site, Muscat, Oman
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Damascus, Syria

REFERENCES:
- [Result] Taher A, Al Jefri A, Elalfy MS, Al Zir K, Daar S, Rofail D, Baladi JF, Habr D, Kriemler-Krahn U, El-Beshlawy A. Improved treatment satisfaction and convenience with deferasirox in iron-overloaded patients with beta-Thalassemia: Results from the ESCALATOR Trial. Acta Haematol. 2010;123(4):220-5. doi: 10.1159/000313447. Epub 2010 Apr 27. PMID 20424435
- See also: Results for CICL670A2402 from the Novartis Clinical Trials website — https://www.ncbi.nlm.nih.gov/pubmed/20424435